CLINICAL TRIAL: NCT03298594
Title: A Specific Cervicograph for Women Attempting at Vaginal Delivery After Cesarean Section: is the Management of Labor Improved?
Brief Title: A Specific Cervicograph for Women Attempting at Vaginal Delivery After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Michel Boulvain, MD, PhD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12-173 MATPED 12-036
Record Dates: First submitted 2017-09-26; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Attempted Vaginal Delivery After a Cesarean Section

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The cervicograph of all participants will be reviewed by two assessors blinded to the study group. In order to be blinded, lines will be added to the cervicographs of the control group by a third party not involved in the evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- specific cervicograph (Experimental): Specific cervicograph, including an alert line (normal progression of cervical dilation, i.e. 1 cm per hour) and an action line 2 hours after the alert line. This should be completed after the diagnose of active labor
  Interventions: Diagnostic Test: specific cervicograph
- Usual cervicograph (No Intervention): The usual cervicograph in our unit is not having lines

INTERVENTIONS:
Diagnostic Test: specific cervicograph
  Other Names: usual cervicograph
  Arms: specific cervicograph

SUMMARY:
The main objective is to evaluate a specific cervicograph (the graph describing the cervical dilation, included in the partograph) for pregnant women with an history of cesarean section, to improve the management of labor for women attempting at a vaginal delivery (VBAC). Women will be randomly assigned to this specific cervicograph (including an action line 2 hours after the alert line), or to the normal cervicograph (no lines). The primary outcome is appropriate detection of dystocia.

DETAILED DESCRIPTION:
Appropriate management of labor is essential to minimize the risk of uterine rupture in case of attempt at vaginal delivery after a cesarean section (VBAC). Dystocia is a known risk factor for uterine rupture during labor in women with previous cesarean section. Some studies have shown that this risk increases after 2 hours at the same cervical dilation during labor. The cervicograph is an important tool to detect dystocia during labor. There is currently no specific cervicograph for pregnant women with a history of cesarean section, and no study evaluated the cervicograph in the monitoring of labor for women with a scarred uterus.

The main objective is to evaluate a specific cervicograph (the graph describing the cervical dilation, included in the partograph) for pregnant women with an history of cesarean section, to improve the management of labor for women attempting at a vaginal delivery (VBAC). Women will be randomly assigned to a specific cervicograph (including an action line 2 hours after the alert line), or to the normal cervicograph (no lines).

The outcomes of this randomized trial are: appropriate detection and management of dystocia; uterine rupture; and success of VBAC.

ELIGIBILITY:
Inclusion Criteria:

* Women in labor, admitted for a VBAC at a gestational age of 37 weeks or more
* Single pregnancy
* Cephalic presentation

Exclusion Criteria:

* More than 1 previous cesarean section
* Multiple pregnancies
* Presentations other than cephalic
* History of low vertical uterotomy, classical or inverted T-shaped
* Past history of myomectomy
* Fetal death
* Fetal anomalies
* Placental anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 135 (Actual)
Dates: Start 2013-02-26 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

PRIMARY OUTCOMES:
Detection of dystocia during labor in women with past history of cesarean section | From inclusion in the study (randomization usually from 2cm) until full cervical dilation.
  Appropriate detection and management of dystocia by identifying women with: no progression of cervical dilation for more than 2 hours during labor; or slow progress, defined as a cervical dilation of less than 2 cm in 4 hours; and immediate decision of cesarean section, to be performed within 30 minutes.

SECONDARY OUTCOMES:
Uterine rupture during labor in women with past history of cesarean section | From inclusion in the study (randomization usually from 2cm) until delivery
  Uterine rupture will be defined as a complete separation of the uterine scar that resulted in protrusion of fetal or placental parts in the peritoneal cavity

OTHER OUTCOMES:
Percentage of VBAC | at delivery
  Percentage of vaginal delivery in women with past history of cesarean section

IPD SHARING:
Plan to Share IPD: No